CLINICAL TRIAL: NCT01759537
Title: Evaluation of Changes of Hard and Soft Tissues After Epi-crestal and Sub-crestal Placement of Ankylos Dental Implants.
Brief Title: Study to Evaluate Bone and Gum Dimension Changes Around Dental Implants Placed in Different Positions in Bone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply International (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ankylos-Bluestone
Record Dates: First submitted 2012-12-31; First posted 2013-01-03 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Mouth, Edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Intervention Model Description: This was a split mouth study design in which the same patient was used for both arms.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implants placed at sub-crestal position. (Experimental): Ankylos dental endosseous implants-Sub-crestal
  Interventions: Device: Ankylos dental endosseous implants-Sub-crestal
- Epi-crestal implants. (Active Comparator): Ankylos dental endosseous implants-Epi-crestal
  Interventions: Device: Ankylos dental endosseous implants-Epi-crestal

INTERVENTIONS:
Device: Ankylos dental endosseous implants-Sub-crestal — Implants placed subcrestally
  Arms: Implants placed at sub-crestal position.
Device: Ankylos dental endosseous implants-Epi-crestal — Implants placed Epi-crestally
  Arms: Epi-crestal implants.

SUMMARY:
The purpose of this study is to test two standard of care techniques of placing dental implants, and to compare how people's bones and gums respond to two different depths at which implants are placed.

DETAILED DESCRIPTION:
The purpose of this study is to test epicrestal and subcrestal placement of dental implants, and to compare how people's bones and gums respond to two different depths at which implants are placed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have read, understood and signed an informed consent form;
2. Subjects must be 18 to 70 years of age;
3. Subjects must be able and willing to follow study procedures and instructions;
4. Subjects must have indication to receive two implants in a bilateral maxillary or mandibular edentulous areas (for at least 4 months post extraction) in areas of pre-molars (first or second) and molars (first or second);
5. Sufficient width and height of bone to place at least 8mm length and any compatible in diameter Ankylos implant;
6. Sufficient vertical clearance to place a single tooth crown replacement;
7. No apical disorder/inflammation at the area of the implant site.

Exclusion Criteria:

1. Subjects participating in other clinical studies within 1 month prior to screening and/or involving therapeutic intervention (either medical or dental) that could affect bone or soft tissue healing;
2. Female subjects who are pregnant or lactating, or who intend to become pregnant during the study period following entrance into the study;
3. Subjects with parafunctional habits;
4. Subjects who have failed to maintain good plaque control;
5. Subjects with any systemic condition like uncontrolled diabetes mellitus, cancer, HIV, disorders that compromise wound healing, chronic high dose steroid therapy, bone metabolic diseases, radiation or other immuno-suppressive therapy which would preclude periodontal surgery;
6. Absence of occlusal stability in centric occlusion;
7. Subjects with the presence of acute infectious lesions in the areas intended for surgery;
8. History within the last 3 months of weekly or more frequent use of smokeless chewing tobacco, pipe or cigar smoking and cigarette smoking (greater than 10 cigarettes per day)
9. Present alcohol or drug abuse;
10. Angulation requirements of the restoration exceeding approximately 15 degrees;
11. Systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration (e.g. calcium channel blocker, dilantin).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Froum, DDS, Principal Investigator — Bluestone Center for Clinical Research
Locations (1):
- Bluestone Center for Clinical Research, New York, New York, United States

REFERENCES:
- See also: Bluestone Clinic at NYU — http://www.bluestonecenter.org/clinical_trials/studydetail.html?id=56

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who fulfilled the inclusion criteria and required two bilateral implants in the pre-molar (first or second) or molar (first or second) region of the maxilla or mandible, ages 18 through 70 years old were eligible to participate in this study. Patient screenings, enrollment, study procedures, and data collection was conducted at the Bluestone Center for Clinical Research (BCCR), New York University (NYU) College of Dentistry, from April 2012 to April 2019.
Pre-assignment Details: Of the 1022 participants who were assessed for eligibility, 974 were excluded as they did not meet the inclusion criteria, did not show for evaluation, or for other reasons. Forty-eight (48) met inclusion criteria and were randomized to treatment.
Units Other Than Participants: implants
Groups:
- Implants Placed at Sub-crestal Position: Ankylos dental endosseous implants placed at sub-crestal position
- Implants Placed at Epi-crestal Position: Ankylos dental endosseous implants placed at epi-crestal position
Period: Overall Study
Arm/Group | Implants Placed at Sub-crestal Position | Implants Placed at Epi-crestal Position
Started | 48; 48 implants (This is a split mouth study. The same 48 patients started the study for both Arms. Three (3) subjects were enrolled but withdrawn and not included in the statistical analysis.) | 48; 48 implants (This is a split mouth study. The same 48 patients started the study for both Arms. Three (3) subjects were enrolled but withdrawn and not included in the statistical analysis.)
Completed | 35; 35 implants (This is a split mouth study. The same 35 patients completed the study for both Arms.) | 35; 35 implants (This is a split mouth study. The same 35 patients completed the study for both Arms.)
Not Completed | 13; 13 implants | 13; 13 implants
Not completed — Death | 1 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Lost to Follow-up | 9 | 9
Not completed — Accident involving jaw fracture | 1 | 1
Not completed — Subcrestal implant too coronal | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Implants Placed at Sub-crestal Position and Epi-crestal Position: Ankylos dental endosseous implants-sub-crestal and epi-crestal
  Ankylos dental endosseous implants-sub-crestal and epi-crestal: Implants placed subcrestally and epi-crestally
Arm/Group | Implants Placed at Sub-crestal Position and Epi-crestal Position
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 21
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Marginal Bone Level (MBL)
Description: Changes in MBLs at 18 months and 30 months after implant placement were chosen as primary outcome parameters. Results are described as mean values and standard deviations.
  Note: Mean changes in MBL for epicrestal and subcrestal placements at lingual and buccal sites is also referred to as "mid-facial bone levels". To determine MBL changes between T0 and each follow-up visit, MBLs at T0 were subtracted from the complementary values for that implant at T18 and T30.
Time Frame: Implant placement, and 18 months and 30 months after implant placement
Population: All subjects available at each time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: implants
Arm/Group | Implants Placed at Sub-crestal Position | Implants Placed at Epi-crestal Position
Number analyzed (Participants) | 43 | 43
Number analyzed (implants) | 43 | 43
mm
  Mean MBL (Buccal) at 18 months after implant placement | -0.14 (0.78) | -0.002 (0.99)
  Mean MBL (Lingual) at 18 months after implant placement | -0.20 (0.59) | -0.07 (0.63)
  Mean MBL (Buccal) at 30 months after implant placement: number analyzed (Participants) | 41 | 41
  Mean MBL (Buccal) at 30 months after implant placement: number analyzed (implants) | 41 | 41
  Mean MBL (Buccal) at 30 months after implant placement | -0.19 (0.99) | 0.36 (0.95)
  Mean MBL (Lingual) at 30 months after implant placement: number analyzed (Participants) | 41 | 41
  Mean MBL (Lingual) at 30 months after implant placement: number analyzed (implants) | 41 | 41
  Mean MBL (Lingual) at 30 months after implant placement | -0.26 (0.57) | 0.27 (0.62)

2. Secondary Outcome: Change in Mid-Buccal Soft Tissue Height
Description: Soft tissue levels were measured clinically from a fixed reference point to the mid buccal soft tissue margin using a stent. Measurements were made from fixed reference points, by using a stent to perform clinical measurements in a reproducible position.
Time Frame: From final restoration (6 months after implant placement), and 12 months, 18 months, 30 months, 42 months, 54 months, and 66 months after implant placement
Population: All subjects available at each time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: implants
Arm/Group | Implants Placed at Sub-crestal Position | Implants Placed at Epi-crestal Position
Number analyzed (Participants) | 43 | 43
Number analyzed (implants) | 43 | 43
mm
  Change in Mid-Buccal Soft Tissue Height at 12 months after implant placement | -0.17 (0.91) | -0.11 (0.76)
  Change in Mid-Buccal Soft Tissue Height at 18 months after implant placement | -0.11 (0.86) | -0.12 (0.78)
  Change in Mid-Buccal Soft Tissue Height at 30 months after implant placement: number analyzed (Participants) | 41 | 41
  Change in Mid-Buccal Soft Tissue Height at 30 months after implant placement: number analyzed (implants) | 41 | 41
  Change in Mid-Buccal Soft Tissue Height at 30 months after implant placement | -0.26 (0.87) | -0.08 (0.81)
  Change in Mid-Buccal Soft Tissue Height at 42 months after implant placement: number analyzed (Participants) | 40 | 40
  Change in Mid-Buccal Soft Tissue Height at 42 months after implant placement: number analyzed (implants) | 40 | 40
  Change in Mid-Buccal Soft Tissue Height at 42 months after implant placement | -0.46 (0.96) | -0.24 (0.85)
  Change in Mid-Buccal Soft Tissue Height at 54 months after implant placement: number analyzed (Participants) | 40 | 40
  Change in Mid-Buccal Soft Tissue Height at 54 months after implant placement: number analyzed (implants) | 40 | 40
  Change in Mid-Buccal Soft Tissue Height at 54 months after implant placement | -0.55 (0.81) | -0.32 (0.96)
  Change in Mid-Buccal Soft Tissue Height at 66 months after implant placement: number analyzed (Participants) | 35 | 35
  Change in Mid-Buccal Soft Tissue Height at 66 months after implant placement: number analyzed (implants) | 35 | 35
  Change in Mid-Buccal Soft Tissue Height at 66 months after implant placement | -0.40 (0.83) | -0.30 (1.14)

3. Secondary Outcome: Change of Interproximal Levels After Final Restoration
Description: Analysis of interproximal bone height change measured by periapical radiographs. The height of the papilla will be assessed at the mesial and distal sites of the implants, by means of the published "papilla Jemt index". Measurements will be assessed by reviewing the clinical photographs.
  Reference: Jemt, T. (1997) "Regeneration of gingival papillae after single-implant treatment". International Journal of Periodontics and Restorative Dentistry 17: 326-333.
Time Frame: From final restoration (6 months after implant placement), and 18 months, 30 months, 42 months, 54 months, and 66 months after implant placement
Population: All subjects available at each time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: implants
Arm/Group | Implants Placed at Sub-crestal Position | Implants Placed at Epi-crestal Position
Number analyzed (Participants) | 43 | 43
Number analyzed (implants) | 43 | 43
mm
  Change in interproximal level at 18 months after implant placement | 0.21 (0.48) | 0.28 (0.46)
  Change in interproximal level at 30 months after implant placement: number analyzed (Participants) | 41 | 41
  Change in interproximal level at 30 months after implant placement: number analyzed (implants) | 41 | 41
  Change in interproximal level at 30 months after implant placement | 0.25 (0.44) | 0.30 (0.44)
  Change in interproximal level at 42 months after implant placement: number analyzed (Participants) | 40 | 40
  Change in interproximal level at 42 months after implant placement: number analyzed (implants) | 40 | 40
  Change in interproximal level at 42 months after implant placement | 0.24 (0.49) | 0.29 (0.50)
  Change in interproximal level at 54 months after implant placement: number analyzed (Participants) | 40 | 40
  Change in interproximal level at 54 months after implant placement: number analyzed (implants) | 40 | 40
  Change in interproximal level at 54 months after implant placement | 0.23 (0.54) | 0.31 (0.55)
  Change in interproximal level at 66 months after implant placement: number analyzed (Participants) | 35 | 35
  Change in interproximal level at 66 months after implant placement: number analyzed (implants) | 35 | 35
  Change in interproximal level at 66 months after implant placement | 0.16 (0.56) | 0.26 (0.64)

4. Secondary Outcome: Change in Marginal Bone Level (MBL)
Description: Changes in MBLs at 66 months after implant placement were chosen as a secondary outcome parameter. Results are described as mean values and standard deviations.
  Note: Mean changes in MBL for epicrestal and subcrestal placements at lingual and buccal sites is also referred to as "mid-facial bone levels". To determine MBL changes between T0 and each follow-up visit, MBLs at T0 were subtracted from the complementary values for that implant at T18, T30 and T66.
Time Frame: Implant placement, and 66 months after implant placement
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: implants
Arm/Group | Implants Placed at Sub-crestal Position | Implants Placed at Epi-crestal Position
Number analyzed (Participants) | 35 | 35
Number analyzed (implants) | 35 | 35
mm
  Mean MBL (Buccal) at 66 months after implant placement | -0.64 (1.66) | -0.30 (2.11)
  Mean MBL (Lingual) at 66 months after implant placement | -0.34 (0.81) | 0.07 (0.74)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from initial implant to 60 months after final restoration
Arm/Group | Implants Placed at Sub-crestal Position | Implants Placed at Epi-crestal Position
All-Cause Mortality (participants affected / at risk) | 1/48 | 1/48
Serious Adverse Events (participants affected / at risk) | 2/48 | 2/48
Other Adverse Events (participants affected / at risk) | 17/48 | 11/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implants Placed at Sub-crestal Position (N=48) | Implants Placed at Epi-crestal Position (N=48)
Death (General disorders) | 1 (1) | 1 (1) — Note: Cause of death is unknown and therefore "General disorders" was selected.
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — An accident involving a fractured upper and lower jaw (trauma adjacent to a study implant)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implants Placed at Sub-crestal Position (N=48) | Implants Placed at Epi-crestal Position (N=48)
Healing abutment lost (Product Issues) | 6 (6) | 2 (2)
Provisional crown loosened/lost (Product Issues) | 3 (3) | 2 (3)
Provisional crown chipped/fractured (Product Issues) | 0 (0) | 1 (1)
Final crown loosened/lost (Product Issues) | 7 (8) | 4 (6)
Final crown chipped/fractured (Product Issues) | 4 (4) | 4 (5)

LIMITATIONS AND CAVEATS:
Several limitations within the present study should be noted with regard to: 1) CT scan performance, 2) intraoral radiograph outcomes, 3) soft tissue level outcomes, 4) periodontal and peri-implant status, and 5) restorative procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less